CLINICAL TRIAL: NCT02493257
Title: Double-Blinded Randomized Prospective Trial of Intranasal Capsaicin Treatment for Non-Allergic Irritant Rhinitis
Brief Title: Intranasal Capsaicin Treatment for Non-Allergic Irritant Rhinitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: American Academy of Otolaryngic Allergy (Other)
Responsible Party: Principal Investigator, Denna Awni Zebda, Associate Professor, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HSC-MS-14-0173
Record Dates: First submitted 2014-11-03; First posted 2015-07-09 (Estimated); Results first posted 2020-08-17 (Actual); Last update posted 2020-08-17 (Actual); Status verified 2020-07

CONDITIONS: Nonallergic Irritant Rhinitis
Keywords: nonallergic irritant rhinitis; nasal congestion; rhinorrhea
MeSH Terms: conditions — Nasal Obstruction; Rhinorrhea | interventions — Capsaicin; Ethanol; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- intranasal capsaicin (Experimental): The capsaicin solution will be prepared by using the formula previously reported by Van Rijswijk et al; (0.1mmol/l) diluted in ethanol and 0.9% normal saline (19). Using the mucosal atomizer device (MAD), 0.8 milliliters (mL) will be delivered to each nasal cavity for a total of 24.4 ug per nasal cavity. 5 consecutive applications of capsaicin or placebo will be administered intranasally, with 1 hour between each application.
  Interventions: Drug: Capsaicin
- Vehicle solution (Placebo Comparator): 100 μL of 1% ethanol in 0.9% saline solution. 5 consecutive applications of capsaicin or placebo will be administered intranasally, with 1 hour between each application.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Capsaicin
  Other Names: intranasal capsaicin
  Arms: intranasal capsaicin
Drug: Placebo
  Other Names: 1% ethanol in 9% saline
  Arms: Vehicle solution

SUMMARY:
The proposed study seeks to investigate the effect of intranasal capsaicin treatment in patient with Non-allergic irritant rhinitis (NAIR), as well as evaluate optical rhinometry (ORM) as a means to quantify symptomatic improvement in NAIR patients during and after treatment.

DETAILED DESCRIPTION:
A study by Lambert et. al. (2012) was able to objectively identify patients with NAIR by intranasal capsaicin challenge followed by assessment with optical rhinometry. Studies have shown that capsaicin therapy can improve symptoms of patients historically identified with NAIR via visual analog scale (VAS) rating of symptoms and symptom surveys; however, there has been no study evaluating the capsaicin therapy on patients objectively identified as NAIR patients.

Multiple studies have demonstrated that intranasal capsaicin can improve nasal symptoms of NAIR patients. Regarding the usage of capsaicin, there is a product on the market: Sinus Buster which has capsaicin as the active ingredient. Numerous research papers have evaluated the efficacy and safety of Sinus Buster for the treatment of congestion in non-allergic rhinitis patients. However, the diagnosis of NAIR in these previous studies was based primarily on history. In addition, the primary outcome in these studies was symptomatic without any objective evaluation. The goal of this study will be two-fold: with patients objectively identified as NAIR patients via the optical rhinometer, we will re-evaluate the therapeutic action of intranasal capsaicin on the management of rhinitic symptoms. We expect that the patients will show significant improvement in their symptoms. We will then use optical rhinometry as a means to objectively monitor changes in symptoms in NAIR patients. We expect that post treatment, patients will no longer have the positive response previously seen on intranasal capsaicin challenge before receiving treatment. We hope to be able to establish optical rhinometry as an objective measurement of symptom improvement for NAIR symptoms, along with the subjective patient surveys.

ELIGIBILITY:
Inclusion criteria:

* Non-allergic irritant rhinitis (NAIR) patients as defined by history (symptoms of nasal congestion, rhinorrhea, nasal itching or sneezing upon exposure to nasal irritants)
* Patients with positive optical rhinometer (ORM) response with intranasal challenge with 0.5 millimolar (mM) capsaicin as described by Lambert et al 2012
* Confirmed negative skin prick test to common allergens (which rules out allergic rhinitis)

Exclusion Criteria:

* History of sinonasal surgery
* Chronic rhinosinusitis
* Inflammatory or granulomatous diseases
* Asthma
* Allergic rhinitis
* Immunocompromised state
* Radiation to the head and neck
* Intranasal steroid use >4 wks
* Intranasal or systemic antihistamine x 3 days
* Intranasal or systemic decongestants x 3 days

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2014-10; Primary Completion 2019-08-02 (Actual); Study Completion 2019-08-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amber U Luong, MD, PhD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Intranasal Capsaicin: The capsaicin solution will be prepared by using the formula previously reported by Van Rijswijk et al; (0.1mmol/l) diluted in ethanol and 0.9% normal saline (19). Using the mucosal atomizer device (MAD), 0.8 millimeters (mL) will be delivered to each nasal cavity for a total of 24.4 ug per nasal cavity. 5 consecutive applications of capsaicin or placebo will be administered intranasally, with 1 hour between each application.
  Capsaicin
- Vehicle Solution: 100 μL of 1% ethanol in 0.9% saline solution. 5 consecutive applications of capsaicin or placebo will be administered intranasally, with 1 hour between each application.
  Placebo
Period: Overall Study
Arm/Group | Intranasal Capsaicin | Vehicle Solution
Started | 11 | 11
4 Week Follow up | 11 | 11
12 Week Follow up | 10 | 10
Completed | 10 | 10
Not Completed | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Intranasal Capsaicin: The capsaicin solution will be prepared by using the formula previously reported by Van Rijswijk et al; (0.1mmol/l) diluted in ethanol and 0.9% normal saline (19). Using the MAD, 0.8 millimeters (0.8mL) will be delivered to each nasal cavity for a total of 24.4 ug per nasal cavity. 5 consecutive applications of capsaicin or placebo will be administered intranasally, with 1 hour between each application.
  Capsaicin
- Total: Total of all reporting groups
Arm/Group | Intranasal Capsaicin | Vehicle Solution | Total
Number analyzed (Participants) | 11 | 11 | 22
Age, Continuous [Mean (Standard Deviation); unit: years] | 40 (16) | 33 (8) | 36.5 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 6 | 9
  Male | 8 | 5 | 13
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  African American | 1 | 1 | 2
  Asian | 1 | 3 | 4
  Caucasian | 8 | 7 | 15
  Hispanic | 1 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 11 | 11 | 22

OUTCOME MEASURES:

1. Primary Outcome: Change in Total Symptom Score
Description: The Total Symptom Score (TSS) uses a visual analog scale (VAS) to assess typical nasal symptoms of non-allergic rhinitis (NAR), including sneezing, nasal irritation, nasal obstruction, and nasal congestion. The TSS is based on a commonly used rhinitis rating system recommended by the FDA for clinical trial studies on non-allergic rhinitis. 4 symptoms (sneezing, nasal irritation, nasal obstruction, and nasal congestion) are rated on a VAS ranging from 0 (none, no distress) to 10 (agonizing, unbearable distress). The TSS total score is the sum of the VAS score for each of the 4 symptoms, with the TSS total score ranging from 0 (none, no distress) to 40 (agonizing, unbearable distress).
Time Frame: baseline and 4 weeks
Measure: Median (Inter-Quartile Range); unit: score on a scale
Groups:
- Intranasal Capsaicin: The capsaicin solution will be prepared by using the formula previously reported by Van Rijswijk et al; (0.1mmol/l) diluted in ethanol and 0.9% normal saline (19). Using the MAD, 0.8mL will be delivered to each nasal cavity for a total of 24.4 ug per nasal cavity. 5 consecutive applications of capsaicin or placebo will be administered intranasally, with 1 hour between each application.
  Capsaicin
Arm/Group | Intranasal Capsaicin | Vehicle Solution
Number analyzed (Participants) | 11 | 11
score on a scale | -5 [-12 to -2] | 2 [-4 to 3]

2. Primary Outcome: Change in Total Symptom Score
Description: as for outcome 1
Time Frame: baseline and 12 weeks
Population: Data was not collected for 1 participant in the intranasal capsaicin arm and 1 participant in the vehicle solution arm.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Intranasal Capsaicin | Vehicle Solution
Number analyzed (Participants) | 10 | 10
score on a scale | -4.5 [-13 to 0] | 1.5 [-2 to 8]

3. Primary Outcome: Change in Nasal Blood Flow as Indicated by Change in Maximal Optical Density Assessed by Optical Rhinometry
Description: Optical rhinometry provides continuous measurement of blood flow in nasal vessels (via optical density measurements), which serves as an indirect assessment of nasal congestion. A greater decrease in optical density (OD) from baseline indicates less nasal blood flow and decreased congestion relative to baseline.
Time Frame: baseline and 4 weeks
Measure: Median (Inter-Quartile Range); unit: log ratio of light in to light out (OD)
Arm/Group | Intranasal Capsaicin | Vehicle Solution
Number analyzed (Participants) | 11 | 11
log ratio of light in to light out (OD) | -0.05 [-0.38 to 0.04] | -0.05 [-0.12 to 0.12]

4. Primary Outcome: Change in Nasal Blood Flow as Indicated by Change in Maximal Optical Density Assessed by Optical Rhinometry
Description: as for outcome 3
Time Frame: baseline and 12 weeks
Population: Data was not collected for one participant in the intranasal capsaicin arm and for one participant in the vehicle solution arm.
Measure: Median (Inter-Quartile Range); unit: log ratio of light in to light out (OD)
Arm/Group | Intranasal Capsaicin | Vehicle Solution
Number analyzed (Participants) | 10 | 10
log ratio of light in to light out (OD) | -0.08 [-0.41 to 0.15] | -0.05 [-0.13 to 0.17]

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | Intranasal Capsaicin | Vehicle Solution
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/11
Other Adverse Events (participants affected / at risk) | 0/11 | 0/11

LIMITATIONS AND CAVEATS:
Small sample size; 2 patients lost to follow-up at 12 weeks; inability to identify NAR patients with elevated local Immunoglobulin E (IgE) levels, which may contribute to limited improvement in some NAR patients in the intervention group.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-11-18): https://cdn.clinicaltrials.gov/large-docs/57/NCT02493257/Prot_SAP_000.pdf